CLINICAL TRIAL: NCT01979263
Title: Attention Bias Modification Treatment for Anxious Youth
Acronym: ABMT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment/data collection
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1207012686R001-IRB
Record Dates: First submitted 2013-09-30; First posted 2013-11-08 (Estimated); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Generalized Anxiety Disorder; Separation Anxiety Disorder; Social Phobia; Specific Phobia; Obsessive-Compulsive Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder; Anxiety, Separation; Phobia, Social; Phobia, Specific; Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Attention Bias Modification (Active Comparator): Attention Bias Modification computer task
  Interventions: Other: Attention Bias Modification Computer Task
- Placebo Computer Task (Placebo Comparator): Placebo computer task
  Interventions: Other: Placebo Computer Task

INTERVENTIONS:
Other: Attention Bias Modification Computer Task — Computer task aimed at actively modifying attention bias
  Arms: Attention Bias Modification
Other: Placebo Computer Task — Computer task that does not actively modify attention bias
  Arms: Placebo Computer Task

SUMMARY:
The purpose of this project is to study the feasibility and efficacy of attention bias modification treatment (ABMT) in a randomized-controlled sample of anxious youth.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether or not ABMT computer-based interventions can be used successfully to help reduce anxiety disorder symptoms in children ages 7 to 17. ABMT is different from most other treatments for anxiety because it is not medication or talk therapy. ABMT is a computerized attention training program designed to change how we direct our attention. The purpose of ABMT is to set in place attentional patterns that do not lead to excessive anxiety. Research has shown that it may be highly effective in reducing anxiety. The Intervention will be composed of your child engaging in 6 brief weekly ABMT sessions. The sessions seem like a repetitive computer game.

This study is appropriate for children who may have symptoms of an anxiety disorder, like Generalized Anxiety Disorder, Separation anxiety Disorder, Social Anxiety Disorder, Specific Phobia, or Obsessive-Compulsive Disorder." Children who appear eligible for the study may attend a diagnostic evaluation and assessment if they meet study criteria.

If a child is eligible for the study, he or she will be randomly assigned to either get an "active" form of the computer program or a "placebo" or inactive form of the computer program. The child will come to six weekly appointments at our clinic that are quite brief, about a half hour. Then the child will have an evaluation after the last of the six appointments to see if the computer intervention was helpful in reducing his or her anxiety. We'd then wait a month and then have a final evaluation to see if the child's anxiety has changed over that period of time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis on Anxiety Disorders Interview Schedule for Diagnostic and Statistical Manual-IV Child and Parent versions of Separation Anxiety Disorder, Social Phobia, Specific Phobia, Obsessive-Compulsive Disorder, or Generalized Anxiety Disorder
* Age 7 to 17

Exclusion Criteria:

* Posttraumatic stress disorder or primary diagnosis of major depressive disorder
* Seizure disorder
* Current treatment with psychotropic medication
* Multiple chronic learning disabilities and/or conduct problems

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2013-10; Primary Completion 2017-01-17 (Actual); Study Completion 2017-01-17 (Actual)

PRIMARY OUTCOMES:
Change in clinical severity ratings on Anxiety Disorder Interview Schedule-Child and Parent Version | after a 6-week intervention and 4-week no-treatment follow-up

SECONDARY OUTCOMES:
Variation in genes associated with treatment response | week 1
  We will study allelic variation in a gene that has been associated with treatment response to anxiety interventions, the serotonin-transporter-linked promoter region (5-HTTLPR)

CONTACTS AND LOCATIONS:
Overall Officials: Megan H Feltenberger, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - Payne Whitney Manhattan Child Division, New York, New York
  - New York Presbyterian Hospital--Westchester Division, White Plains, New York

IPD SHARING:
Plan to Share IPD: Yes